CLINICAL TRIAL: NCT00174421
Title: Genotropin in Short Children Born Small for Gestational Ag - A Long-Term Study in Belgium
Brief Title: Treatment Of Short Stature With Genotropin In Children Born Small For Gestational Age Until Final Height
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-8122-011; A6281219
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Growth Disorder
MeSH Terms: conditions — Growth Disorders | interventions — Therapeutics; Human Growth Hormone

INTERVENTIONS:
Drug: Treatment with Genotropin in different dosages

SUMMARY:
This trial evaluates whether long-term treatment with Genotropin normalizes final (adult) height in short children born small for gestational age

ELIGIBILITY:
Inclusion Criteria:

* Participation in the 90-080 study

Exclusion Criteria:

* Any severe, acute or chronic disease
* Any other identifiable reason for short stature

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 2001-04; Study Completion 2005-08

PRIMARY OUTCOMES:
Final height, compared to the expected familial target height

SECONDARY OUTCOMES:
Body weight, body mass index at final height; adverse events and assessment of hematological and clinical chemistry

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer